CLINICAL TRIAL: NCT01127581
Title: Phase III, Double-blind, Randomized, Multicenter Study of Exogenous Prostaglandin Comparing the Efficacy & Safety of the MVI 200 mcg Versus the Dinoprostone Vaginal Insert (DVI) for Reducing Time to Vaginal Delivery in Pregnant Women at Term
Brief Title: Efficacy & Safety Study Comparing Misoprostol Vaginal Insert (MVI) Versus Dinoprostone Vaginal Insert (DVI) for Reducing Time to Vaginal Delivery
Acronym: EXPEDITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Miso-Obs-303
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Reducing Time to Vaginal Delivery; Cervical Ripening; Induction of Labor
Keywords: Misoprostol vaginal insert; Dinoprostone vaginal insert; Cervidil; Cervical ripening; Induction of labor; Rate of cesarean section
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MVI 200 (Experimental): MVI 200 mcg vaginal insert
  Interventions: Drug: MVI 200
- Dinoprostone Vaginal Insert (DVI) (Active Comparator): 10 mg Dinoprostone vaginal insert
  Interventions: Drug: Dinoprostone Vaginal Insert (DVI)

INTERVENTIONS:
Drug: MVI 200 — Dose reservoir of 200 mcg of misoprostol in a hydrogel polymer vaginal insert within a retrieval system. The MVI 200 will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
  Other Names: Misopess(TM); Misodel (R)
  Arms: MVI 200
Drug: Dinoprostone Vaginal Insert (DVI) — Dose reservoir of 10 mg of dinoprostone in a hydrogel polymer vaginal insert within a retrieval system. The DVI will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
  Other Names: Cervidil (R); Propess (R)
  Arms: Dinoprostone Vaginal Insert (DVI)

SUMMARY:
The purpose of this study is to determine whether the Misoprostol Vaginal Insert (MVI) 200 microgram (mcg) can decrease the time to vaginal delivery compared to the Dinoprostone Vaginal Insert (DVI) 10 milligram (mg) in pregnant women requiring cervical ripening and induction of labor.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Pregnant women at ≥ 36 weeks 0 days inclusive gestation;
* Women aged 18 years or older;
* Candidate for pharmacological induction of labor;
* Single, live vertex fetus;
* Baseline modified Bishop score ≤ 4;
* Parity ≤ 3 (parity is defined as one or more births live or dead after 24 weeks gestation);
* Body Mass Index (BMI) ≤ 50 at the time of entry to the study.

Exclusion Criteria:

* Women in active labor;
* Presence of uterine or cervical scar or uterine abnormality e.g., bicornate uterus. Biopsies, including cone biopsy of the cervix, are permitted;
* Administration of oxytocin or any cervical ripening or labor inducing agents (including mechanical methods) or a tocolytic drug within 7 days prior to enrollment. Magnesium sulfate is permitted if prescribed as treatment for pre-eclampsia or gestational hypertension;
* Severe pre-eclampsia marked by Hemolytic anemia, Elevated Liver enzymes, Low Platelet count (HELLP) syndrome, other end-organ affliction or Central Nervous System (CNS) findings other than mild headache;
* Fetal malpresentation;
* Diagnosed congenital anomalies, not including polydactyly;
* Any evidence of fetal compromise at baseline (e.g., non-reassuring fetal heart rate pattern or meconium staining);
* Amnioinfusion or other treatment of non-reassuring fetal status at any time prior to the induction attempt;
* Ruptured membranes ≥ 48 hours prior to the start of treatment;
* Suspected chorioamnionitis;
* Fever (oral or aural temperature > 37.5°C);
* Any condition in which vaginal delivery is contraindicated e.g., placenta previa or any unexplained genital bleeding at any time after 24 weeks during this pregnancy;
* Known or suspected allergy to misoprostol, dinoprostone, other prostaglandins or any of the excipients;
* Any condition urgently requiring delivery;
* Unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1358 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (34):
- United States (34):
  - Maricopa Medical Center - District Medical Group, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Phoenix Perinatal Associates (Scottsdale Healthcare Shea), Scottsdale, Arizona
  - Watching Over Mothers and Babies Foundation, Tucson, Arizona
  - Miller's Childrens Hospital, Long Beach, California
  - UCI Medical Center, Orange, California
  - The Women's Clinic of Northern Colorado, Fort Collins, Colorado
  - Christiana Care Health System (DE Center for MFM), Newark, Delaware
  - University of FL College of Medicine, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas School of Medicine, Kansas City, Kansas
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - St. Louis University, St Louis, Missouri
  - St. Peters University Hospital, New Brunswick, New Jersey
  - University of New Mexico/New Mexico Health Science Center, Albuquerque, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Brody School of Medicine, Greenville, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Clinical Trials of America, Eugene, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University Medical Group/Greenville Hospital System, Greenville, South Carolina
  - UT College of Medicine Chattanooga, Erlanger Health System, Chattanooga, Tennessee
  - High Risk Obstetrical Consultants, PLLC, Knoxville, Tennessee
  - Research Memphis Associates, Memphis, Tennessee
  - University of Texas Health Sciences Center at Houston, Houston, Texas
  - Salt Lake Women's Center, PC, Sandy City, Utah
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Derived] Miller H, Goetzl L, Wing DA, Powers B, Rugarn O. Optimising daytime deliveries when inducing labour using prostaglandin vaginal inserts. J Matern Fetal Neonatal Med. 2016;29(4):517-22. doi: 10.3109/14767058.2015.1011117. Epub 2015 Mar 16. PMID 25758619
- [Derived] Wing DA, Brown R, Plante LA, Miller H, Rugarn O, Powers BL. Misoprostol vaginal insert and time to vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2013 Aug;122(2 Pt 1):201-209. doi: 10.1097/AOG.0b013e31829a2dd6. PMID 23857539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women who required to be induced were recruited at 35 sites in the US.
Groups:
- Dinoprostone Vaginal Insert (DVI): 10 mg Dinoprostone vaginal insert
  Dinoprostone vaginal insert: Dose reservoir of 10 mg of dinoprostone in a hydrogel polymer vaginal insert within a retrieval system. The DVI will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
Period: Overall Study
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Started | 678 | 680
Completed | 678 | 680
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI) | Total
Number analyzed (Participants) | 678 | 680 | 1358
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 678 | 680 | 1358
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.99) | 25.9 (5.95) | 26.0 (5.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 678 | 680 | 1358
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 678 | 680 | 1358

OUTCOME MEASURES:

1. Primary Outcome: Time to Vaginal Delivery During the First Hospital Admission
Time Frame: Interval from study drug administration to vaginal delivery (average 24 hours)
Population: Subjects who underwent a cesarean delivery during the first hospitalization were censored using the longest time interval from study drug administration to cesarean delivery, independent of treatment assignment. Subjects who were discharged prior to delivery or withdrew consent prior to delivery were also censored.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
minutes | 1292.00 [1200.00 to 1402.00] | 1968.50 [1812.00 to 2093.00]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Subjects who underwent a cesarean delivery during the first hospitalization were censored using the longest time interval from study drug administration to cesarean delivery during the first hospitalization, independent of treatment group. Subjects who, in their first hospitalization, were discharged prior to delivery or withdrew consent prior to delivery were censored using the longest time interval from study drug administration to labor and delivery discharge, independent of treatment group; Test type: Superiority or Other; p < 0.001, Log Rank; Median Difference (Net) = -677 — Sample size 675 per group provides 90% power to see an improvement of ≥320 minutes (20% improvement from DVI) in time to vaginal delivery between MVI 200 & DVI assuming a median time of 1600 minutes for DVI & 34% dropout rate based on 5% 2-sided test

2. Primary Outcome: Incidence of Cesarean Delivery During the First Hospital Admission
Time Frame: Interval from study drug administration to cesarean delivery (average 24 hours)
Population: Analysis was based on a between-treatment-group difference in the safety population. Subjects discharged prior to delivery, withdrew early without having a cesarean delivery or were lost-to-follow up were classified as not having the event.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
percentage of participants | 25.96 [22.70 to 29.43] | 27.06 [23.75 to 30.57]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); The analysis of the cesarean delivery rates during the first hospitalization was based on a between-treatment-group difference. If the upper limit of the asymptotic two-sided 95% confidence interval of the difference in event rates (MVI minus DVI) was less than the calculated non-inferiority margin (10% relative to the DVI rate, i.e., 0.1 times DVI rate), then MVI 200 would be considered non-inferior to DVI; Test type: Non-Inferiority or Equivalence — A sample size of 675 subjects per group will provide a sufficient number of subjects to assess non-inferiority of MVI 200 with respect to rate of cesarean delivery, based on an alpha level of 5% and 80% power for a two-sided approach using a 10% non-inferiority limit (relative to the DVI rate), assuming a 30% rate of cesarean delivery in the DVI group compared to a 26% rate in the MVI 200 group; Chi-squared; Difference in Populations = -1.10, 95% CI 2-sided [-5.79 to 3.59] — MVI 200 - DVI

3. Secondary Outcome: Time to Any Delivery (Vaginal or Cesarean) During the First Hospital Admission
Time Frame: Interval from study drug administration to neonate delivery (average 24 hours)
Population: Subjects who did not deliver during the first hospitalization were censored at the time of labour and delivery discharge.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
minutes | 1096.50 [1031.00 to 1170.00] | 1639.50 [1573.00 to 1731.00]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Subjects who did not deliver during the first hospitalization were censored using the longest time interval from study drug administration to labor and delivery discharge without delivery, independent of treatment group; Test type: Superiority or Other; p < 0.001, Log Rank; Median Difference (Net) = -543 — MVI 200 - DVI

4. Secondary Outcome: Time to Active Labor During the First Hospital Admission
Description: Active labor was defined as progressive cervical dilatation to 4 cm with any frequency of contractions OR rhythmic, firm, adequate quality uterine contractions causing progressive cervical change occurring at a frequency of 3 or more in 10 minutes and lasting 45 seconds or more.
Time Frame: Interval from study drug administration to active labor (average 12 hours)
Population: Intention-to-Treat (ITT) population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
minutes | 726.50 [719.00 to 773.00] | 1116.50 [1083.00 to 1352.00]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Subjects who never went into active labor during the first hospitalization were censored using the longest time interval from study drug administration to delivery during the first hospitalization, independent of treatment group. Subjects who, in their first hospitalization, were discharged prior to delivery or withdrew consent prior to delivery were censored using the longest time interval from study drug administration to labor and delivery discharge, independent of treatment group; Test type: Superiority or Other; p < 0.001, Log Rank; Median Difference (Net) = -390 — MVI 200 - DVI

5. Secondary Outcome: Incidence of Pre-delivery Oxytocin During the First Hospital Admission
Description: Percentage of participants in receipt of Oxytocin for induction after study drug removal.
Time Frame: At least 30 minutes after study drug removal
Population: Analysis population includes subjects who delivered during the first hospitalization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 674 | 671
percentage of participants | 48.1 [44.24 to 51.92] | 74.1 [70.58 to 77.35]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = -26 — MVI 200 - DVI

6. Secondary Outcome: Incidence of Vaginal Delivery Within 12 Hours
Time Frame: Interval from study drug administration to vaginal delivery within 12 hours
Population: Intention-to-Treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
percentage of participants | 19.76 [16.83 to 22.96] | 8.38 [6.41 to 10.72]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 9.67 — MVI 200 - DVI

7. Secondary Outcome: Incidence of Any Delivery Within 24 Hours
Time Frame: Interval from study drug administration to delivery of neonate within 24 hours
Population: Intention-to-Treat (ITT) Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
percentage of participants | 67.70 [64.03 to 71.21] | 40.74 [37.02 to 44.54]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 26.96 — MVI 200 - DVI

8. Secondary Outcome: Incidence of Any Delivery Within 12 Hours
Time Frame: Interval from study drug administration to delivery of neonate within 12 hours
Population: Intention-to-Treat (ITT) Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
percentage of participants | 23.16 [20.03 to 26.52] | 9.26 [7.19 to 11.70]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 13.90 — MVI 200 - DVI

9. Secondary Outcome: Incidence of Vaginal Delivery Within 24 Hours
Time Frame: Interval from study drug administration to vaginal delivery within 24 hours
Population: Intention-to-Treat (ITT) Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
percentage of participants | 54.57 [50.74 to 58.37] | 33.97 [30.41 to 37.67]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 29.80 — MVI 200 - DVI

10. Secondary Outcome: Incidence of Vaginal Delivery
Time Frame: Interval from study drug administration to vaginal delivery (average 24 hours)
Population: The Intention-to-Treat (ITT) population was used for all secondary efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
percentage of participants | 73.30 [69.80 to 76.60] | 71.62 [68.07 to 74.98]
Statistical Analysis 1: Comparison: MVI 200 vs Dinoprostone Vaginal Insert (DVI); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 1.68 — MVI 200 - DVI

11. Secondary Outcome: Rate of Adverse Events
Description: All adverse events were rated by the Investigator as mild, moderate or severe and classified as having no relationship, possible relationship or a probable relationship to the study drug.
Time Frame: From study drug administration to hospital discharge (approximately 48-72 hours)
Population: The percentage of subjects with adverse events are presented for the Intrapartum (before delivery), postpartum (maternal) and neonatal periods.
Measure: Number; unit: percentage of participants
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Number analyzed (Participants) | 678 | 680
percentage of participants
  Subjects with an Intrapartum Adverse Events | 55.5 | 54.6
  Subjects with Maternal Postpartum Adverse Events | 21.4 | 21.2
  Subjects with Neonatal Adverse Events | 53.4 | 58.1

ADVERSE EVENTS:
Time Frame: All adverse events were followed until resolution or at least 30 days after discontinuation of the study drug, whichever occurred first.
Description: All adverse events occurring to the maternal-fetal unit (pre-delivery/ intrapartum), the mother (postpartum) or the neonate were recorded. Adverse events that resulted in a cesarean delivery were reported as serious adverse events as they were medically significant events that routinely prolonged the duration of hospitalization.
Arm/Group | MVI 200 | Dinoprostone Vaginal Insert (DVI)
Serious Adverse Events (participants affected / at risk) | 130/678 | 107/680
Other Adverse Events (participants affected / at risk) | 520/678 | 533/680
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVI 200 (N=678) | Dinoprostone Vaginal Insert (DVI) (N=680)
Disseminated intravascular coagulation # (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — # Postpartum Event
Polycythaemia * (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — * Neonatal Event
Pericarditis # (Cardiac disorders) | 0 (0) | 1 (1) — # Postpartum Event
Supraventricular tachycardia * (Cardiac disorders) | 1 (1) | 0 (0) — * Neonatal Event
Supraventricular tachycardia + (Cardiac disorders) | 0 (0) | 1 (1) — + Intrapartum Event
Adrenogenital syndrome * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — * Neonatal Event
Anal atresia * (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — * Neonatal Event
Ankyloglossia congenital * (Congenital, familial and genetic disorders) | 3 (3) | 2 (2) — * Neonatal Event
Anomalous pulmonary venous connection * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — * Neonatal Event
Atrial septal defect * (Congenital, familial and genetic disorders) | 8 (8) | 6 (6) — * Neonatal Event
Cataract congenital * (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — * Neonatal Event
Congenital choroid plexus cyst * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — * Neonatal Event
Congenital hydronephrosis * (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — * Neonatal Event
Congenital nose malformation * (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — * Neonatal Event
Congenital pyelocaliectasis * (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) — * Neonatal Event
Cryptorchism * (Congenital, familial and genetic disorders) | 6 (6) | 2 (2) — * Neonatal Event
Hydrocele * (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) — * Neonatal Event
Hypospadias * (Congenital, familial and genetic disorders) | 4 (4) | 4 (4) — * Neonatal Event
Patent ductus arteriosus * (Congenital, familial and genetic disorders) | 4 (4) | 4 (4) — * Neonatal Event
Penile torsion * (Congenital, familial and genetic disorders) | 3 (3) | 1 (1) — * Neonatal Event
Phimosis * (Congenital, familial and genetic disorders) | 0 (0) | 3 (3) — * Neonatal Event
Pilonidal cyst congenital * (Congenital, familial and genetic disorders) | 3 (3) | 7 (7) — * Neonatal Event
Polydactyly * (Congenital, familial and genetic disorders) | 3 (3) | 3 (3) — * Neonatal Event
Pulmonary artery stenosis congenital * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — * Neonatal Event
Supernumerary nipple * (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) — * Neonatal Event
Syndactyly * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — * Neonatal Event
Talipes * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — * Neonatal Event
VACTERL syndrome * (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) — * Neonatal Event
Ventricular septal defect * (Congenital, familial and genetic disorders) | 4 (4) | 1 (1) — * Neonatal Event
Vitreous haemorrhage * (Eye disorders) | 0 (0) | 1 (1) — * Neonatal Event
Anal fistula * (Gastrointestinal disorders) | 0 (0) | 1 (1) — * Neonatal Event
Intestinal obstruction * (Gastrointestinal disorders) | 1 (1) | 0 (0) — * Neonatal Event
Salivary gland enlargement * (Gastrointestinal disorders) | 1 (1) | 0 (0) — * Neonatal Event
Fever neonatal * (General disorders) | 1 (1) | 0 (0) — * Neonatal Event
Endometritis # (Infections and infestations) | 2 (2) | 1 (1) — # Postpartum Event
Pneumonia * (Infections and infestations) | 0 (0) | 1 (1) — * Neonatal Event
Pneumonia # (Infections and infestations) | 0 (0) | 1 (1) — # Postpartum Event
Postpartum sepsis # (Infections and infestations) | 1 (1) | 0 (0) — # Postpartum Event
Sepsis neonatal * (Infections and infestations) | 1 (1) | 1 (1) — * Neonatal Event
Septic shock * (Infections and infestations) | 0 (0) | 1 (1) — * Neonatal Event
Skull fracture * (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — * Neonatal Event
Urine output decreased * (Investigations) | 1 (1) | 1 (1) — * Neonatal Event
Feeding disorder neonatal * (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — * Neonatal Event
Joint crepitation * (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — * Neonatal Event
Muscular weakness # (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — # Postpartum Event
Dysaesthesia # (Nervous system disorders) | 1 (1) | 0 (0) — # Postpartum Event
Encephalopathy neonatal * (Nervous system disorders) | 0 (0) | 1 (1) — * Neonatal Event
Hypoxic-ischaemic encephalopathy * (Nervous system disorders) | 4 (4) | 0 (0) — * Neonatal Event
Paraesthesia # (Nervous system disorders) | 0 (0) | 1 (1) — # Postpartum Event
Abnormal labour affecting foetus + (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 0 (0) — + Intrapartum Event
Drug withdrawal syndrome neonatal * (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — * Neonatal Event
Erb's palsy * (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — * Neonatal Event
Foetal acidosis * (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — * Neonatal Event
Foetal heart rate disorder + (Pregnancy, puerperium and perinatal conditions) | 65 (65) | 46 (46) — + Intrapartum Event
Hypoglycaemia neonatal * (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) — * Neonatal Event
Neonatal disorder * (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — * Neonatal Event
Postpartum haemorrhage # (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) — # Postpartum Event
Premature separation of placenta + (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — + Intrapartum Event
Puerperal pyrexia # (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — # Postpartum Event
Retained placenta or membranes # (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — # Postpartum Event
Uterine contractions abnormal + (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — + Intrapartum Event
Uterine rupture + (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — + Intrapartum Event
Weight decrease neonatal * (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — * Neonatal Event
Anxiety # (Psychiatric disorders) | 0 (0) | 1 (1) — # Postpartum Event
Hydronephrosis * (Renal and urinary disorders) | 0 (0) | 1 (1) — * Neonatal Event
Chordee * (Reproductive system and breast disorders) | 1 (1) | 0 (0) — * Neonatal Event
Testicular torsion * (Reproductive system and breast disorders) | 0 (0) | 1 (1) — * Neonatal Event
Vulval haematoma # (Reproductive system and breast disorders) | 0 (0) | 1 (1) — # Postpartum Event
Neonatal aspiration * (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — * Neonatal Event
Neonatal respiratory depression * (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — * Neonatal Event
Neonatal respiratory distress syndrome * (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — * Neonatal Event
Pneumothorax * (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — * Neonatal Event
Transient tachypnoea of the newborn * (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — * Neonatal Event
Deep vein thrombosis # (Vascular disorders) | 1 (1) | 0 (0) — # Postpartum Event
Hypertension # (Vascular disorders) | 1 (1) | 1 (1) — # Postpartum Event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVI 200 (N=678) | Dinoprostone Vaginal Insert (DVI) (N=680)
Abnormal labour affecting foetus + (Pregnancy, puerperium and perinatal conditions) | 59 (62) | 19 (19) — + Intrapartum Event
Arrested labour + (Pregnancy, puerperium and perinatal conditions) | 96 (96) | 128 (129) — + Intrapartum Event
Caput succedaneum * (Pregnancy, puerperium and perinatal conditions) | 58 (58) | 60 (60) — * Neonatal Event
Chorioamnionitis + (Pregnancy, puerperium and perinatal conditions) | 38 (38) | 59 (59) — + Intrapartum Event
Foetal heart rate disorder + (Pregnancy, puerperium and perinatal conditions) | 124 (138) | 138 (160) — + Intrapartum Event
Hyperbilirubinaemia neonatal * (Pregnancy, puerperium and perinatal conditions) | 62 (62) | 78 (78) — * Neonatal Event
Meconium in amniotic fluid + (Pregnancy, puerperium and perinatal conditions) | 120 (120) | 92 (92) — + Intrapartum Event
Postpartum haemorrhage # (Pregnancy, puerperium and perinatal conditions) | 40 (41) | 37 (37) — # Postpartum Event
Umbilical cord around neck * (Pregnancy, puerperium and perinatal conditions) | 184 (184) | 194 (194) — * Neonatal Event
Neonatal respiratory depression * (Respiratory, thoracic and mediastinal disorders) | 34 (34) | 30 (30) — * Neonatal Event
Infection prophylaxis * (Surgical and medical procedures) | 46 (46) | 63 (63) — * Neonatal Event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any abstract,presentation or manuscript proposed for publication must be submitted to the Sponsor for review at least 30 days prior to submission for any meeting or journal.If deemed necessary by the Sponsor for protection of proprietary information prior to patent filing,the Investigator agrees to a further delay of 60 days before any presentation or publication is submitted.Publications must be in a form that does not reveal technical information that is considered confidential or proprietary.